CLINICAL TRIAL: NCT00631592
Title: GSK1349572 Repeat Dose Escalation Study
Brief Title: GSK1349572 Repeat Dose Escalation and Relative Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ING111322
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2010-10

CONDITIONS: Healthy Subjects
Keywords: GSK1349572,; healthy volunteers,; repeat dose,; relative bioavailability; Healthy subjects
MeSH Terms: interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSK1349572 (Other): GSK1349572
  Interventions: Drug: GSK1349572

INTERVENTIONS:
Drug: GSK1349572

SUMMARY:
This is a repeat dose escalation study of GSK1349572 followed by a relative bioavailability study comparing tablet and suspension formulations in healthy volunteers.

DETAILED DESCRIPTION:
ING111322: A Double-Blind, Randomized, Placebo-Controlled, Repeat Dose Escalation Study to Investigate the Safety, Tolerability and Pharmacokinetics of GSK1349572 Followed by A Single Dose, Randomized, 3-Period, Balanced, Crossover Study to Assess the Relative Bioavailability of Two Formulations and Food Effect on GSK1349572 in Healthy Male and Female Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 50 years of age.
* A female subject is eligible to participate if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any female who:

  * Is pre-menopausal with a documented bilateral tubal ligation, bilateral oophorectomy (removal of the ovaries) or hysterectomy, or
  * Is post-menopausal defined as 12 months of spontaneous amenorrhea. A follicle stimulating hormone (FSH) level will be performed to confirm a post-menopausal status. For this study, FSH levels > 40 mlU/ml is confirmatory. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt, HRT should be discontinued for 2 weeks and then the subject rescreened, as HRT can suppress FSH.
* Male subjects must agree to use one of the contraception methods listed in protocol. This criterion must be followed from the time of the first dose of study medication until 14 days after the last dose of study medication.
* Body weight >/ 50 kg for men and >/ 45 kg for women and BMI within the range 18.5-31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as:
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* If heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* Has a history or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy should be excluded.
* screening ECG within protocol parameters (a single repeat is allowed for eligibility determination):• Evidence of previous myocardial infarction (Does not include ST segment changes associated with repolarization).
* Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], WPW syndrome).
* Sinus Pauses > 3 seconds.
* Any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety for the individual subject.
* Non-sustained or sustained ventricular tachycardia (3 consecutive ventricular ectopic beats).
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting surgery or percutaneous transluminal coronary angioplasty or any clinically significant cardiac disease.
* History/evidence of clinically significant pulmonary disease.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), direct bilirubin or creatinine values greater than the upper limit of normal. A single repeat is allowed for eligibility determination.
* History of significant renal or hepatic diseases.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2008-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
adverse events; clinical hematology, clinical chemistry, urinalysis, vital signs (blood pressure and heart rate), electrocardiogram (ECG) intervals, ECG rhythm, and ECG axis from predose values, pharmacokinetic parameters throughout the study | throughout the study

SECONDARY OUTCOMES:
Pre-morning dose concentrations (Ct) on Day 2 through 10 to assess the achievement of steady state of GSK1349572 following repeat administration. | day 2 thru day10
Day 10 AUC(0-t), Cmax, C0, Ct, and Cmin following last repeat dose administration at different doses for the assessment of dose proportionality. | day 10
Single dose plasma GSK1349572 pharmacokinetic parameters: tmax, t1/2, tlag and CL/F. | single dose
pharmacokinetic parameters | throughout the study
Plasma AUC(0-t) and AUC(0-¥) of midazolam, with and without GSK1349572 co-administration (Day -1 and Day 10). | Day -1 and Day 10

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No